CLINICAL TRIAL: NCT03585543
Title: Self-Management for Youth and Families Living With Sickle Cell Disease - SMYLS
Brief Title: Self-Management for Youth and Families Living With SCD - SMYLS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: Pro00062837
Record Dates: First submitted 2018-05-04; First posted 2018-07-13 (Actual); Results first posted 2020-04-16 (Actual); Last update posted 2020-11-19 (Actual); Status verified 2020-10

CONDITIONS: Sickle Cell Disease
MeSH Terms: conditions — Anemia, Sickle Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single group intervention arm (Experimental)
  Interventions: Behavioral: Voice Crisis Alert V2

INTERVENTIONS:
Behavioral: Voice Crisis Alert V2 — Intervention consists of a mHealth app delivered via smartphone

SUMMARY:
The purpose of this proposal is to integrate family-centered self-management strategies with mobile health (mHealth) technology to improve reach, self-management behaviors, and child and caregiver physical and psychosocial symptoms and quality of life. Specifically, the investigators propose to conduct feasibility testing of SMYLS, which has been adapted based on user feedback in the first phase of this study. First the investigators will work with the Medical University of South Carolina (MUSC) Pediatric Sickle Cell Clinic to identify and recruit families with children with sickle cell disease (SCD) in the community, statewide. Next, the investigators will test the feasibility of the intervention with 30 dyads of children ages 8 - 17 with sickle cell disease and their parent or primary caregiver, (N=60)

ELIGIBILITY:
Inclusion Criteria:

* children ages 8 - 17 years and parent or primary caregiver 18 years or older
* child with sickle cell disease, as reported by clinician at MUSC Pediatric Sickle Cell Clinic

Exclusion Criteria:

* Parent/caregiver or child with cognitive disability or delay that precludes ability to participate
* Lack of wi-fi access

Ages: 8 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Actual)
Dates: Start 2018-03-16 (Actual); Primary Completion 2019-01-31 (Actual); Study Completion 2019-01-31 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Group Receiving mHealth Intervention: This was a single-arm study; all participants received the intervention.
Period: Overall Study
Arm/Group | Group Receiving mHealth Intervention
Started | 30
Mid-intervention Assessment (6-weeks) | 25
End-of-intervention Assessment (12 Weeks | 22
3-month Post-intervention Follow-up (6 m | 15
Completed | 15
Not Completed | 15

BASELINE CHARACTERISTICS:
Groups:
- Intervention Group: This was a single-arm study; all participants received the intervention.
Arm/Group | Intervention Group
Number analyzed (Participants) | 30
Age, Continuous [Mean (Standard Deviation); unit: years] | 11.8 (2.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14
  Male | 16
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 30
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 30
  White | 0
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 30
Parent/caregiver type [Count of Participants; unit: Participants]
  mother | 27
  father | 1
  grandmother | 2
Parent/caregiver employment status [Count of Participants; unit: Participants]
  employed | 21
  caregiver/stay-at-home parent | 2
  unemployed | 3
  student | 0
  disabled | 0
  unknown/no response | 4
Parent/caregiver education level [Count of Participants; unit: Participants]
  9 - 12 grade or less | 3
  high school graduate or GED | 5
  some college or certification course | 13
  college graduate or above | 9
Parent/caregiver marital status [Count of Participants; unit: Participants]
  married | 9
  living with partner | 1
  single | 17
  divorced | 3
household size [Mean (Standard Deviation); unit: number of people] | 3.4 (1.5)

OUTCOME MEASURES:

1. Primary Outcome: Rates of Recruitment
Description: Number of weeks required to recruit 30 participants.
Time Frame: Assessed each week over a period of 6 months, cumulative data up to 6 months is reported.
Measure: Number; unit: weeks
Arm/Group | Intervention Group
Number analyzed (Participants) | 30
weeks | 14

2. Primary Outcome: Participant Adherence to Intervention
Description: Number of participants who used the intervention (mHealth application) from baseline to mid-intervention, from mid-intervention to end-of-intervention, and from end-of-intervention to follow-up, assessed by number of participants who logged into and used the app, stored in the app's back end database.
Time Frame: baseline to 6 weeks, 6 weeks to 12 weeks, 12 weeks to 6 months
Measure: Number; unit: participants
Arm/Group | Intervention Group
Number analyzed (Participants) | 30
participants
  Number who used from baseline to 6 weeks | 30
  Number who used from 6 weeks to 12 weeks | 15
  Number who used from 12 weeks to 6 months | 10

3. Primary Outcome: Acceptability of Intervention
Description: Number of participants reporting problems with the intervention (mHealth app) per week.
Time Frame: Assessed each week over a period of 6 months, cumulative data up to 6 months is reported.
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention Group
Number analyzed (Participants) | 30
Participants | 4

4. Primary Outcome: Participant Adherence to Intervention
Description: number of participants who accessed the educational component of intervention, assessed using back end app use database
Time Frame: baseline to 6 weeks, 6 weeks to 12 weeks, 12 weeks to 6 months
Measure: Number; unit: participants
Arm/Group | Intervention Group
Number analyzed (Participants) | 30
participants
  Number who used from baseline to 6 weeks | 28
  Number who used from 6 weeks to 12 weeks | 7
  Number who used from 12 weeks to 6 months | 4

5. Primary Outcome: Participant Adherence to Intervention
Description: Number of participants who accessed the symptom monitoring component of the intervention, assessed using the app back end database
Time Frame: baseline to 6 weeks, 6 weeks to 12 weeks, 12 weeks to 6 months
Measure: Number; unit: participants
Arm/Group | Intervention Group
Number analyzed (Participants) | 30
participants
  Number who used from baseline to 6 weeks | 29
  Number who used from 6 weeks to 12 weeks | 15
  Number who used from 12 weeks to 6 months | 10

6. Primary Outcome: Participant Adherence to Intervention
Description: number of participants who sent messages to nurse practitioner
Time Frame: baseline to 6 weeks, 6 weeks to 12 weeks, 12 weeks to 6 months
Measure: Number; unit: participants
Arm/Group | Intervention Group
Number analyzed (Participants) | 30
participants
  Number who used from baseline to 6 weeks | 12
  Number who used from 6 weeks to 12 weeks | 2
  Number who used from 12 weeks to 6 months | 1

7. Secondary Outcome: Difference in Mean Pain Score Rating From Baseline to End-of-intervention
Description: Patient Reported Outcome Measurement Information System (PROMIS) Pain Interference Pediatric Short Form 8a: Change in score at 12 weeks minus baseline. Raw scores range from 0 - 32, with 0 being the lowest pain rating and 32 the highest pain rating. Any decrease in mean difference between scores = improved
Time Frame: baseline, 12 weeks
Population: 20 participants retained to 12 weeks (end-of-intervention) for analysis
Measure: Mean (95% Confidence Interval); unit: scores on scale
Arm/Group | Group Receiving mHealth Intervention
Number analyzed (Participants) | 20
scores on scale | -9.0 [-15.0 to -3.0]

8. Secondary Outcome: Difference in Mean Caregiver Self-efficacy Score From Baseline to End-of-intervention
Description: Self-efficacy for Managing Chronic Disease 6-item scale. Scores for each item range from 1 - 10 with 1 indicating lower confidence/self-efficacy and 10 indicating higher confidence/self-efficacy. Scores for each item are averaged for the mean total score. Change in score at 12 weeks minus baseline. Any increase in difference in mean scores = improved
Time Frame: baseline, 12 weeks
Population: 20 participants retained to 12 weeks
Measure: Mean (95% Confidence Interval); unit: scores on scale
Arm/Group | Group Receiving mHealth Intervention
Number analyzed (Participants) | 20
scores on scale | 0.2 [-0.5 to 0.9]

9. Secondary Outcome: Differences in Mean Scores for Quality of Life From Baseline to End-of-intervention
Description: Pediatric Quality of Life Inventory (Peds QL): Scores are transformed on a scale from 0 - 100, with 0 indicating the highest possible problems with quality of life and 100 indicating the lowest possible problems with quality of life. Change in score at 12 weeks minus baseline. Any increase in difference between mean scores = improved
Time Frame: baseline, 12 weeks
Population: 20 participants retained to end-of-intervention for analysis
Measure: Mean (95% Confidence Interval); unit: scores on scale
Arm/Group | Group Receiving mHealth Intervention
Number analyzed (Participants) | 20
scores on scale | 10.9 [4.3 to 17.4]

10. Secondary Outcome: Difference in Mean Scores for Fatigue From Baseline to End-of-intervention
Description: Patient Reported Outcomes Measurement Information System (PROMIS) Fatigue Pediatric Short Form 10a: Raw Scores range from 0 - 40 with 0 being the least amount of fatigue and 40 the most fatigue. Difference in mean scores at 12 weeks minus baseline. Any decrease in rating = improved
Time Frame: baseline, 12 weeks
Population: 20 participants retained to end-of-intervention for analysis
Measure: Mean (95% Confidence Interval); unit: scores on scale
Arm/Group | Group Receiving mHealth Intervention
Number analyzed (Participants) | 20
scores on scale | -7.9 [-12.9 to -2.9]

11. Secondary Outcome: Difference in Mean Scores for Anxiety From Baseline to End-of-intervention
Description: Patient Reported Outcomes Measurement System (PROMIS) Pediatric Short Form Anxiety 8a: Raw Scores range from 0 - 32, with 0 being the lowest anxiety rating and 32 the highest anxiety rating. Change in score at 12 weeks minus baseline. Any decrease difference in mean scores = improved
Time Frame: baseline, 12 weeks
Population: 20 participants retained to end-of-intervention for analysis
Measure: Mean (95% Confidence Interval); unit: scores on scale
Arm/Group | Group Receiving mHealth Intervention
Number analyzed (Participants) | 20
scores on scale | 1.6 [-3.7 to 6.8]

12. Secondary Outcome: Differences in Mean Scores on Depressive Symptoms From Baseline to End-of-intervention
Description: Patient Reported Outcomes Measurement System (PROMIS) Pediatric short form depression 8a: Raw Scores range from 0 - 32, with 0 being the lowest depression rating and 32 the highest depression rating. Change in score at 12 weeks minus baseline. Any decrease in differences in mean scores = improved
Time Frame: baseline,12 weeks
Population: 20 participants retained to end-of-intervention for analysis
Measure: Mean (95% Confidence Interval); unit: scores on scale
Arm/Group | Group Receiving mHealth Intervention
Number analyzed (Participants) | 20
scores on scale | -3.1 [-7.3 to 1.1]

13. Secondary Outcome: Differences in Mean Scores for Pain Intensity From Baseline to End-of-intervention
Description: Patient Reported Outcome Measurement Information System (PROMIS) Pain Intensity Pediatric 3a. Raw scores range from 3 - 15, with 3 being the lowest pain intensity rating and 15 being the highest pain intensity rating. Change in score at 12 weeks minus baseline. Any decrease in mean difference between scores = improved
Time Frame: baseline, 12 weeks
Population: 20 participants retained to end-of-intervention
Measure: Mean (95% Confidence Interval); unit: scores on scale
Arm/Group | Group Receiving mHealth Intervention
Number analyzed (Participants) | 20
scores on scale | -1.9 [-4.4 to 0.6]

14. Secondary Outcome: Differences in Mean Scores for Disease-related Quality of Life From Baseline to End-of-intervention
Description: Pediatric Quality of Life Inventory (Peds QL) with SCD module: Scores are transformed on a scale from 0 - 100, with 0 indicating the highest possible problems with quality of life and 100 indicating the lowest possible problems with quality of life. Change in score at 12 weeks minus baseline. Any increase in difference between mean scores = improved
Time Frame: baseline, 12 weeks
Population: 20 participants retained to end-of-intervention for analysis
Measure: Mean (95% Confidence Interval); unit: scores on scale
Arm/Group | Group Receiving mHealth Intervention
Number analyzed (Participants) | 20
scores on scale | 12.5 [7.1 to 17.9]

15. Secondary Outcome: Clinic Appointment Attendance
Description: Number of missed clinic appointments at baseline compared to 12 weeks
Time Frame: 12 weeks
Population: Limitations of this feasibility study included issues with the wording and participant interpretation of clinic appointment attendance questions, leading to an inability to accurately assess clinic appointment attendance.
Arm/Group | Intervention Group
Number analyzed (Participants) | 0

16. Secondary Outcome: Home Medication Administration
Description: Adherence to home medications, measured by number of medications marked as taken in the app database.
Time Frame: 12 weeks
Population: Limitations of this feasibility study included technical difficulties with the app, leading to an inability to accurately assess home medication administration.
Arm/Group | Intervention Group
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: The duration of study participation; 6 months
Arm/Group | Intervention Group
All-Cause Mortality (participants affected / at risk) | 0/30
Serious Adverse Events (participants affected / at risk) | 2/30
Other Adverse Events (participants affected / at risk) | 0/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intervention Group (N=30)
Vaso-occlusive crisis (Blood and lymphatic system disorders) | 2 (2) — Participants were hospitalized for occurrence of vaso-occlusive crisis

LIMITATIONS AND CAVEATS:
Limitations of this feasibility study included technical difficulties with the app, leading to an inability to accurately assess medication adherence data and measurement issues with the clinic appointment attendance. We were unable to assess these additional outcome measures with accuracy.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-09-25): https://cdn.clinicaltrials.gov/large-docs/43/NCT03585543/Prot_SAP_000.pdf
  • Informed Consent Form (2017-08-28): https://cdn.clinicaltrials.gov/large-docs/43/NCT03585543/ICF_001.pdf